CLINICAL TRIAL: NCT05302856
Title: CMV IGG Antibodies in Semen as a Predictor for Blood Testis Barrier Damage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Chana Adler, Principal Investigator, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IGGSEMEN-HMO-CTIL
Record Dates: First submitted 2022-02-28; First posted 2022-03-31 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Male Infertility
Keywords: sperm; blood testis barrier; cmv antibody; unexplained infertility
MeSH Terms: conditions — Infertility, Male | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Presumably fertile male patients going through ART treatment (Experimental)
  Interventions: Diagnostic Test: Blood test (CMV IGG, Anti sperm antibody, Testosterone levels)
- Subfertile/infertile male patients with abnormal semen analysis (Experimental)
  Interventions: Diagnostic Test: Blood test (CMV IGG, Anti sperm antibody, Testosterone levels)
- Male patients suffering from unexplained infertility (Experimental)
  Interventions: Diagnostic Test: Blood test (CMV IGG, Anti sperm antibody, Testosterone levels)

INTERVENTIONS:
Diagnostic Test: Blood test (CMV IGG, Anti sperm antibody, Testosterone levels) — Peripheric blood extraction

SUMMARY:
To assess whether the presence of Cytomegalovirus (CMV) Immunoglobulin G (IGG) antibodies in semen is a reliable predictor of male subfertility or infertility.

DETAILED DESCRIPTION:
Prospective cohort study performed in the artificial reproductive technology (ART) unit.

The study will evaluate semen and serum samples from the following groups:

1. Presumably fertile male patients going through ART treatment (for preimplantation genetic testing (PGT) or female indications).
2. Subfertile/infertile male patients with abnormal semen analysis.
3. Male patients suffering from unexplained infertility. All samples will be collected on the day of ovum retrieval procedure, and the semen samples will be evaluated only after completing the fertilization process. The samples will be tested for CMV IGG antibodies and testosterone levels in semen and serum. In addition, anti-sperm antibodies will be measured in the serum. The ratio between CMV IGG antibodies in semen and serum will be calculated, and will be compared with presence of hormone profile, semen analysis parameters and ART parameters.

ELIGIBILITY:
Inclusion Criteria:

* All male patients addressing the infertility unit in Hadassah Mt Scopus for IVF procedure

Exclusion Criteria:

* Refusal to participate
* Male partner utilizing pre cycle frozen sperm sample
* Donor sperm cycles
* Surgically retrieved sperm

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
CMV antibody ratio serum/semen | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Haverfield JT, Meachem SJ, Nicholls PK, Rainczuk KE, Simpson ER, Stanton PG. Differential permeability of the blood-testis barrier during reinitiation of spermatogenesis in adult male rats. Endocrinology. 2014 Mar;155(3):1131-44. doi: 10.1210/en.2013-1878. Epub 2013 Jan 1. PMID 24424039
- [Background] Stanton PG. Regulation of the blood-testis barrier. Semin Cell Dev Biol. 2016 Nov;59:166-173. doi: 10.1016/j.semcdb.2016.06.018. Epub 2016 Jun 25. PMID 27353840